CLINICAL TRIAL: NCT06768359
Title: The Effect of Manual Acupuncture and Standard Therapy on Anxiety and Quality of Life Scores in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Deity Indrayati Nugraha, Medical doctor, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 24-12-1826
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Quality of Life; Cancer
MeSH Terms: conditions — Anxiety Disorders; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The manual acupuncture and standard therapy will be designed as the intervention group, while the sham acupuncture and standard therapy will be designed as the control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants, and outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The manual acupuncture and standard therapy
  Interventions: Procedure: Manual acupuncture and standard therapy
- Control Group (Sham Comparator): The sham acupuncture and standard therapy
  Interventions: Procedure: Sham acupuncture and standard therapy

INTERVENTIONS:
Procedure: Manual acupuncture and standard therapy — Manual acupuncture is acupuncture needle insertion was done perpendicularly to the acupuncture points GV20, EXHN3, HT7, and PC6 using Huanqiu needle measuring 0.25 x 25mm with mild stimulation rotation technique at a speed of 60x/minute and needle retention for 30 minutes. Therapy was performed every day for 6 days.
  Standard therapy is anxiolytic drugs and supportive psychotherapy given to patients according to the decision of the psychiatrist treating the patient.
  Arms: Intervention Group
Procedure: Sham acupuncture and standard therapy — Sham acupuncture is when acupuncture needles are inserted into acupuncture points, but do not actually penetrate the skin, only attached to the plaster. Therapy was performed every day for 6 days.
  Standard therapy is anxiolytic drugs and supportive psychotherapy given to patients according to the decision of the psychiatrist treating the patient.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to prove that the combination of acupuncture therapy and standard therapy is more effective in reducing anxiety and improving the quality of life of cancer patients. The main questions it aims to answer are:

1. Can the combination of manual acupuncture and standard therapy reduce anxiety based on Hamilton Anxiety Rating Scale (HAM-A) scores in cancer patients compared to the sham acupuncture and standard therapy group?
2. Can the combination of manual acupuncture and standard therapy improve the quality of life of cancer patients based on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC-QLQ C30) compared to the sham acupuncture and standard therapy group?

Participants will:

Get manual acupuncture therapy and also standard therapy, such as oral Benzodiazepin and supportive psychotherapy or sham acupuncture therapy and the standard therapy (Benzodiazepin and supportive psychotherapy) every day for 6 days.

Researchers will compare the changes of anxiety scores and quality of life between cancer patients who received manual acupuncture therapy and standard therapy, and cancer patients who received sham acupuncture and standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-59 years.
* Diagnosed with cancer in the last 6 months
* Experiencing moderate to severe anxiety (assessed by HAM-A Score > 14)
* Willing to participate in this study until completion and sign an informed consent.

Exclusion Criteria:

* Cancer patients with unstable hemodynamics
* Cancer patients with brain metastases
* Patients who have been diagnosed with anxiety disorders and have received pharmacological therapy from psychiatrists before.
* Patients who have contraindications to manual acupuncture (there are wounds or infections at the point to be punctured, patients are allergic to stainless steel, patients are phobic of needles)
* Patients who are uncooperative and do not allow acupuncture therapy (patients who are restless, angry)
* Patients with poor liver function (SGOT (Serum Glutamic Oxaloacetic Transaminase) /SGPT (serum glutamate pyruvate transaminase)values increase 2-3 times the normal value)
* Patients with blood clotting disorders (platelets <50,000, INR (International Normalized Ratio) > 2)
* Patients with neutropenia (Absolute neutrophil count <1000)
* Patients with overt DIC (disseminated intravascular coagulation) and acute venous or arterial thrombosis

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Hamilton anxiety rating scale (HAM-A) score | 6 days
  One tool to measure the degree of anxiety symptoms is a questionnaire. Scores range from 0-56.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC-QLQ C30) score | 6 days
  Questionnaire to assess the quality of life of cancer patients with anxiety. Scores range from 0-100

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee of Faculty of Medicine; KEPK RS Kanker Dharmais, Principal Investigator — The Health Research Ethics Commitee of Dharmais Cancer Hospital
Locations (2):
- Indonesia (2):
  - Universitas Indonesia, Jakarta Pusat, DKI Jakarta
  - RS Kanker Dharmais, Jakarta

IPD SHARING:
Plan to Share IPD: No